CLINICAL TRIAL: NCT02319512
Title: Effects of Chewing Gum Against Postoperative Ileus After Pancreaticoduodenectomy - a Randomized Controlled Trial
Brief Title: Effects of Chewing Gum Against Postoperative Ileus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a radical change in postoperative care as well as surgical technique.
Sponsor: Thomas Andersson (Other)
Responsible Party: Sponsor-Investigator, Thomas Andersson, RN, CNS, MSc, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1818111; VGFOUGSB-1818111 (Other Grant/Funding Number: Research and Development in Sweden)
Record Dates: First submitted 2014-12-07; First posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Chewing Gum; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chewing gum (Experimental): Chewing gum was administered every fourth hour (08.00-12.00, 12.00-16.00 and 16.00-20.00). During each four-hour period, patients chewed two pieces of gum for 30 minutes each. Chewing gum was used during the whole hospital stay.
  Interventions: Other: Chewing gum
- Control (Sham Comparator): Controls received standard care and sips of glucose, in total 3.6g/day in a 12-ml mixture per day, the same amount of glucose per day as the treatment group received via the chewing gum
  Interventions: Other: Glucose

INTERVENTIONS:
Other: Chewing gum — ChiczaTM organic chewing gum 6 pieces a day
  Arms: Chewing gum
Other: Glucose — 12ml glucose solution (13,6g) per day
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether the use of chewing gum effects postoperative ileus after pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Postoperative ileus is common after surgery. One non-pharmacological intervention that has shown promising results in reducing the duration of postoperative ileus is chewing gum after surgery. However, this has not been investigated in upper gastrointestinal surgery such as pancreatic surgery. Hence the aim of this study was to investigate the effects of chewing gum treatment on patients undergoing pancreaticoduodenectomy due to pancreatic or periampullary cancer.

This study was conducted as a phase-III trial. Patients diagnosed with pancreatic tumours scheduled for pancreaticoduodenectomy were included. The treatment group received chewing gum postoperatively and standard care. Controls received glucose solution and standard care.

Participants were included on the day of admission, which was the day prior to surgery. Randomization to the two groups (1:1) was done when patients returned from the intensive care unit (ICU) to the ward. This procedure was chosen in order to avoid perioperative drop-outs due to inoperable tumors. With a power of 80% and a level of significance of 0.05, 18 patients were needed in each group.Comparisons between the groups were analyzed with non-parametric tests; the Mann Whitney U test and Chi 2 test.

Controls received standard care and sips of glucose, in total 3.6g/day in a 12-ml mixture per day, the same amount of glucose per day as the treatment group received via the chewing gum. The chewing gum used was ChiczaTM, a natural organic gum whose main ingredients are latex, glucose and natural flavors (lime or spearmint). Patients started to chew after they returned from the ICU the day after surgery. Chewing gum was administered every fourth hour (08.00-12.00, 12.00-16.00 and 16.00-20.00). During each four-hour period, patients chewed two pieces of gum for 30 minutes each. Chewing gum was used during the whole hospital stay. The time to the first postoperative flatulence and defecation was recorded, in addition to standard clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with pancreatic or periampullary cancer and scheduled to undergo pancreaticoduodenectomy.
* Understand and speak swedish
* No diagnosed neurological injuries or diseases affecting the ability to swallow or gastric function
* No ongoing treatment for mental disease
* No ongoing abuse of alcohol or other drugs
* No previously known allergies to the content of chewing gum

Exclusion Criteria:

* Additional surgery after primary surgery.
* No radical curative surgery
* Previous abdominal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
First flatus after surgery | From day of surgery until first postoperative flatus (with in the first 21 days)
First stool after surgery | From day of surgery until first stool (with in the first 21 days)

SECONDARY OUTCOMES:
Start of clear fluids | From day of surgery until start of clear liquids after surgery (with in the first 21 days)
Start of liquid diet | From day of surgery until start of liquid diet after surgery (with in the first 21 days)
Length of hospital stay | From day of surgery until discharge from surgical ward (with in the first 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Falk, PhD, Study Director — Institute of Health and Care Sciences, Sahlgrenska Academy at Gothenburg University, Gothenburg, Sweden; Monika Fagevik Olsén, PhD, Study Director — Department of Gastrosurgical Research and Education, Sahlgrenska Academy at Gothenburg University, Gothenburg, Sweden; Kristofer Bjerså, PhD, Principal Investigator — Division of Nursing, Department of Neurobiology, Care Sciences and Society, Karolinska Institutet, Stockholm, Sweden; Thomas Andersson, MSc, Principal Investigator — Department of Surgery, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Andersson T, Bjersa K, Falk K, Olsen MF. Effects of chewing gum against postoperative ileus after pancreaticoduodenectomy--a randomized controlled trial. BMC Res Notes. 2015 Feb 10;8:37. doi: 10.1186/s13104-015-0996-0. PMID 25886536